CLINICAL TRIAL: NCT01839695
Title: Valiant Mona LSA Stent Graft System Early Feasibility Study
Brief Title: Safety and Efficacy of Valiant Mona LSA Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10086370DOCRev1C
Record Dates: First submitted 2013-04-11; First posted 2013-04-25 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Thoracic Aortic Aneurysms
Keywords: Thoracic Aneurysm; Endovascular Aortic Repair; TEVAR
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valiant Mona LSA Stent Graft System (Experimental): TEVAR procedure using Medtronic Stent Graft
  Interventions: Device: Valiant Mona LSA Stent Graft System

INTERVENTIONS:
Device: Valiant Mona LSA Stent Graft System — All subjects will be implanted with this device

SUMMARY:
The Valiant Mona LSA thoracic stent graft system is for the endovascular repair of aneurysms of the descending thoracic aorta (DTA) in patients who require coverage of the left subclavian artery (LSA).The study is intended to assess safety and performance of the device acutely and at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* The subject or legal guardian understands the nature of the study and agrees to its provisions on a written informed consent form
* Subject must be considered a candidate for revascularization of the LSA.
* Subject has a DTA which will require coverage of the LSA
* Subject's anatomy must meet the anatomical criteria to receive that implanted device

Exclusion Criteria:

* Subject has had previous endovascular repair of the ascending and/or descending thoracic aorta.
* Subject is in acute renal failure or has renal insufficiency with a serum creatinine ≥ 2.0 mg/dL
* Subject is a pregnant female.
* Enrollment in another clinical study
* Subject has had a cerebral vascular accident (CVA)or myocardial infarction (MI) within 3 months.
* Subject has a history of bleeding diathesis, coagulopathy, or refuses blood transfusion.
* Subject has a known allergy or intolerance to the device components.
* Subject has a known hypersensitivity or contraindication to anticoagulants or contrast media, which is not amenable to pre-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Roselli, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (2):
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- St George's Vascular Institute, St. George's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Roselli EE, Arko FR 3rd, Thompson MM; Valiant Mona LSA Trial Investigators. Results of the Valiant Mona LSA early feasibility study for descending thoracic aneurysms. J Vasc Surg. 2015 Dec;62(6):1465-71.e3. doi: 10.1016/j.jvs.2015.07.078. Epub 2015 Oct 23. PMID 26483004

RESULTS

PARTICIPANT FLOW:
Groups:
- Valiant Mona LSA Stent Graft System: TEVAR procedure using Medtronic Stent Graft>
  > Valiant Mona LSA Stent Graft System: All subjects will be implanted with this device
Period: Overall Study
Arm/Group | Valiant Mona LSA Stent Graft System
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Valiant Mona LSA Stent Graft System
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.89 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 7
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Observation - Rate of Major Adverse Events (MAEs)
Description: Major Adverse Events is a composite endpoint that includes Aneurysm Related Mortality (ARM), Stroke, Paraplegia, and Left Arm/Hand Ischemia.
Time Frame: 1 month
Population: Includes active subjects in the ITT population at 30 days post-index procedure.
Measure: Number; unit: participants
Groups:
- Valiant Mona LSA Stent Graft System: TEVAR procedure using Medtronic Stent Graft >
  > Valiant Mona LSA Stent Graft System: All subjects will be implanted with this device
Arm/Group | Valiant Mona LSA Stent Graft System
Number analyzed (Participants) | 9
participants | 3

2. Primary Outcome: Primary Effectiveness Observation
Description: Treatment success which is defined as technical success (successful delivery and deployment of the stent graft in the planned location with no unintentional coverage of other vessels, assessed intraoperatively, and the removal of the delivery system) and successful exclusion of the aneurysm while maintaining patency of the MSG and BSG at the 30 day visit.
Time Frame: 1 month
Population: Based on the number of ITT subject with evaluable data, subjects were considered unevaluable for treatment success if the 30 day imaging was unable to assess patency of the MSG and BSG. One subject completed CT imaging at discharge, which was not repeated at the 30 day visit, and, therefore, was not considered evaluable for this assessment.
Measure: Number; unit: participants
Arm/Group | Valiant Mona LSA Stent Graft System
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Time Frame: Through 30 days
Description: Investigators are required to assess for adverse events at each follow-up timepoint, including discharge, 30 days, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months. Per protocol, all adverse events are required to be reported, regardless of relationship.
Arm/Group | Valiant Mona LSA Stent Graft System
Serious Adverse Events (participants affected / at risk) | 7/9
Other Adverse Events (participants affected / at risk) | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valiant Mona LSA Stent Graft System (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1)
Cardiovascular Deconditioning (Cardiac disorders) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Cerebellar Infarction (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 2 (2)
Hemianopia (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valiant Mona LSA Stent Graft System (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No